CLINICAL TRIAL: NCT01607281
Title: The Ability of Anesthesiologists Identifying Internal Jugular Vein by Anatomic Landmark Technique
Brief Title: The Ability of Anesthesiologists Identifying Internal Jugular Vein Bilaterally by Anatomic Landmarks
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, derya özkan, md consultant of anesthesiology, Diskapi Teaching and Research Hospital
Other Study IDs: DiskapiTRH1; DiskapiTRH232012 (Registry Identifier: USGIJV232012); USGIJV062012 (Registry Identifier: DiskapiTRH062012)
Record Dates: First submitted 2012-05-18; First posted 2012-05-30 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2012-05

CONDITIONS: Internal Jugular Vein Canulation; Anatomical Landmark
Keywords: anatomical landmark; internal jugular vein canulation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- anesthesiologists, experience: There is one arm. All participating anesthesiologists wıll fulfill the questionary survey and show the imaginary puncture site by USG bilaterally.

SUMMARY:
The study is designed to determine anaesthetists ability to locate the right internal jugular vein(IJV) and left IJV using a landmark technique. Initially, a questionnaire was completed detecting previous user experience. An ultrasound probe, using the midpoint as an 'imaginary needle', was placed on the neck of a healthy volunteer and the image recorded. Both anaesthetist and volunteer were blinded to the screen until the image was stored. Anaesthetists were grouped into senior or junior by the total number of IJV canulation experience. The success rate is going to be measured as pass or fail.

DETAILED DESCRIPTION:
Anesthesiologists are usually qualified in internal jugular vein canulation by using anatomic landmark technique. The anatomy of right IJV and left IJV may differ each other. The hypothesis is that the anatomical difference between right and left IJV may give rise to false puncture of especially left IJV by using anatomical landmark technique.Although USG is available, most of the experienced anesthesiologist does not prefer to use USG for IJV canulation due to different reasons.In addition to this anesthesiologists are generally preferring right IJV canulation, thus they are inexperienced in left IJV canulation. So especially during left IJV canulation,not by anatomical landmark technique but by USG will be recommended for anesthesiologists.

ELIGIBILITY:
Inclusion Criteria:

* The voluntary anesthesiologists who are studying in diskapi training and research hospital

Exclusion Criteria:

* The anesthesiologists who are not willing to participate, the anesthesiologists whom refused to fulfill the questionnaire form.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the residents of anesthesiology clinics
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
determine the difference between anesthesiologists ability to show left and right internal jugular vein by usg probe (pass/fail) | participants will be followed for the duration of operating room stay, an expected average of 15 minutes
  The participants are going to be graded pass/fail according to whether the midline trajectory of the usg probe intersected any part of the lumen of the internal jugular vein. The participating anesthesiologists will show imaginary puncture site for IJV cannulation bilaterally by ultrasonography. The blind investigator will save the ultrasonographic images as jpeg files and another investigator will consider the images.

SECONDARY OUTCOMES:
determine the difference between senior and junior anesthesiologists ability to show left and right internal jugular vein by usg probe (pass/fail). | participants will be followed for the duration of operating room stay, an expected average of 15 minutes
  The participants are going to fulfill a survey asking their experience about IJV canulation. After the survey the anesthesiologists are going to classified as senior/junior. The participants are going to be graded pass/fail according to whether the midline trajectory of the usg probe intersected any part of the lumen of the internal juguler vein.

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of health diskapi yildirim beyazit training and research hospital, Ankara, Altindag, Turkey (Türkiye)

REFERENCES:
- [Background] Harber CR, Harvey DJ, Wiles MD, Bogod DG. The ability of anaesthetists to identify the position of the right internal jugular vein correctly using anatomical landmarks. Anaesthesia. 2010 Sep;65(9):885-8. doi: 10.1111/j.1365-2044.2010.06426.x. PMID 21198484
- [Background] Sulek CA, Blas ML, Lobato EB. A randomized study of left versus right internal jugular vein cannulation in adults. J Clin Anesth. 2000 Mar;12(2):142-5. doi: 10.1016/s0952-8180(00)00129-x. PMID 10818329
- [Background] Muralidhar K. Left internal versus right internal jugular vein access to central venous circulation using the Seldinger technique. J Cardiothorac Vasc Anesth. 1995 Feb;9(1):115-6. doi: 10.1016/s1053-0770(05)80084-9. No abstract available. PMID 7718748